CLINICAL TRIAL: NCT00287768
Title: A Phase III Study of Docetaxel and S-1 Versus S-1 in the Treatment of Advanced Gastric Cancer
Brief Title: Phase III Study of Docetaxel + S-1 vs. S-1 for Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Cancer Research Organization (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Masashi Fujii / Associate Professor, Department of Surgery, Surugadai Nippon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JACCRO GC-03
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; advanced gastric cancer; S-1; docetaxel; phase III study
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Docetaxel + S-1
  Interventions: Drug: docetaxel + S-1
- 2 (Active Comparator): S-1
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: docetaxel + S-1 — Docetaxel iv on day one and S-1 po days 1 to 14 every 3 weeks
  Other Names: taxotere; TS-1
  Arms: 1
Drug: S-1 — S-1 po days 1-28 every 6 weeks
  Other Names: TS-1
  Arms: 2

SUMMARY:
The primary objective of this study is to compare median overall survival of the test arm (docetaxel and S-1) to the control arm (S-1 only) in subjects with advanced or recurrent gastric cancer.

DETAILED DESCRIPTION:
Seven-hundred and fifty thousand of new gastric cancer cases are diagnosed worldwide per year. Advanced gastric cancer (AGC) is considered nearly incurable with less than 10% of subjects alive 5 years after diagnosis. Therefore, new treatment regimens are needed for subjects with AGC.

S-1, a new oral fluoropyrimidine which consists of the 5-FU prodrug tegafur (ftorafur, FT) and two enzyme inhibitors, CDHP (5-chloro-2,4-dihydroxypyridine) and OXO (potassium oxonate), in a molar ratio of 1(FT):0.4 (CDHP):1(OXO) is commercially available since late 90'in Japan. Phase II trials have demonstrated that S-1 is active, as a single agent, for the treatment of gastric (RR 44.6%), colorectal (RR 37.4%), head and neck, breast, non-small cell lung, and pancreatic cancers. In gastric cancer, phase III trials (JCOG 9912) comparing 5-FU alone and CPT-11/CDDP combination are currently underway and these results are awaited. Despite of JCOG 9912 study is ongoing, 80% of patients of AGC are already treated by S-1, because of high RR and convenience use for out-patient basis. P-II studies S-1/CDDP, S-1/CPT-11 and S-1/Docetaxel showed high RR(55-76%) and long MST(12-14M). Furthermore, P-III studies are already conducted S-1 vs. S-1/CDDP and S-1 vs. S-1/CPT-11 in Japan. The aim of this study is to compare S-1/Docetaxel vs. S-1 alone in the patients of AGC. This study is a prospective, multicenter, multinational, non-blinded, randomized phase III study.

Patients: Inoperable or relapse gastric cancer. Informed consent must be obtained in writing before treatment. Subjects meeting all of the inclusion criteria and exclusion criteria will be considered for enrollment into study. Then patients will be randomly assigned into two groups S-1/Docetaxel(Treatment Arm A) or S-1 alone(Treatment Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven in operable advanced gastric adenocarcinoma (including adenocarcinoma of the gastrooesophageal junction) or relapse gastric adenocarcinoma
* Subjects must be able to take orally
* Measurable lesion and/or non-measurable lesion defined by RECIST
* ECOG performance status ≦ 1
* Hgb ≧ 8g/dL, WBC 4000-12000/mm3, platelets ≧ 100,000/mm3
* Creatine ≦ upper normal limit (UNL)
* Total bilirubin ≦ 1.5 X UNL
* AST, ALT and ALP ≦ 2.5 x UNL
* No prior chemotherapy
* Life expectancy estimated than 3 months
* Written informed consent

Exclusion Criteria:

* Active double cancer
* Gastrointestinal bleeding
* Excessive amounts of ascites require drainage
* Known brain metastases
* Symptomatic peripheral neuropathy ≧ garde 2. by NCI-CTCAE ver.3.0
* Pulmonary fibrosis, Intestinal pneumonitis
* History of hypersensitivity to fluoropyrimidines, docetaxel or medications formulated with polysorbate 80
* Any previous chemotherapy or radiotherapy for AGC
* Pregnancy or lactation women, or women with suspected pregnancy or men with willing to get pregnant
* Treatment with any investigational product during the last 4 weeks prior to study entry
* Definite contraindications for the use of corticosteroids
* Any subject judged by the investigator to be unfit for any reason to participate in the study

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
overall survival | median

SECONDARY OUTCOMES:
time-to-progression | From onset of regression to progression
response rate | response during observation
safety | side effects during observation

CONTACTS AND LOCATIONS:
Overall Officials: Masashi Fujii, MD PhD, Principal Investigator — Surugadai Nihon University Hospital
Locations (116):
- Japan (116):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Aichi Medical University Hospital, Okazaki, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Nakadoori General Hospital, Akita, Akita
  - Aomori Prefectural Central Hospital, Aomori, Aomori
  - Hirosahi University Graduate School of Medicine, Hirosaki, Aomori
  - Hirosaki Unuversity,School of Medicine, Hirosaki, Aomori
  - Misawa City Hospital, Misawa, Aomori
  - Department of frontier surgery Graduate school of medicine,Chiba University, Chiba, Chiba
  - Department of Organ kegulatory Surgery (First Department Surgery),Ehime University Graduate School of Medicine, Ehime, Ehime
  - Matsuyama Simin Hospital, Matsuyama, Ehime
  - Fukui Prefectural Hospital, Fukui-shi, Fukui
  - Fukui Red Cross Hospital, Fukui-shi, Fukui
  - Saiseikai Hospital, Fukui-shi, Fukui
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - National Kyusyu Cancer Center, Fukuoka, Fukuoka
  - Kyusyu University Faculty of Medical Sciences, Fukuoka, Fukuoka
  - Kyusyu Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuoka, Fukuoka
  - Iizuka Hospital, Iizuka, Fukuoka
  - Nippon Steel Yawata Memorial Hospital, Kitakyushu, Fukuoka
  - Universsity of Occupational and Environmental Health,Japan, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu Municipal Hospital, Gifu, Gifu
  - Gifu University School of Medicine, Gifu, Gifu
  - Gifu Prefectural Gifu Hospital, Gifu, Gifu
  - Ibi Kose Hospital, Ibi, Gifu
  - Gunma University Hospital, Maehashi, Gunma
  - Gunma Prefectural Cancer Center, Oota, Gunma
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - Horoshima City Asa Hospital, Hiroshima, Hiroshima
  - Hiroshima University Research Institute for Radiation Biology and Medicine Tumor Surgery, Hiroshima, Hiroshima
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Asahikawa-Kosei General Hospital, Asahikawa, Hokkaido
  - Asahikawa Medical College Hospital, Asahikawa, Hokkaido
  - Hakodate Goryoukaku Hopsital, Hakodate, Hokkaido
  - Kushiro City General Hospital, Kushiro, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kinki Central Hospital, Itami, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Hyogo College Of Medicine, Nishimiya, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaragi
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical School Hospital, Kanazawa, Ishikawa-ken
  - Kanazawa Medical University Hospital, Nakajima, Ishikawa-ken
  - Keiju Medical Center, Nanao, Ishikawa-ken
  - Iwate Medical University Hospital, Morioka, Iwate
  - Morioka Red Cross Hospital, Morioka, Iwate
  - Department of surgical oncology and digestive surgery kagoshima university graduate school, Kagoshima, Kagoshima-ken
  - Tokai Medical University Hospital, Isehara, Kanagawa
  - St.Marianna University School of Medicine, Kawasaki, Kanagawa
  - Kitasato University East Hospital, Sagamihara, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Yokohama Citizen's Municipal Hospital, Yokohama, Kanagawa
  - St. Marianna University School of Medicine,Yokohama City Seibu Hospital, Yokohama, Kanagawa
  - Kanagawa Prefectural Cancer Center, Yokohama, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kochi Health Sciences Center, Kochi, Kochi
  - Kumamoto Medical University Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - University Hospital,Kyoto Prefectural University of Medicien, Kyoto, Kyoto
  - Tohoku Rosai Hospital, Sendai, Miyagi
  - Institute of Development,Aging and Cancer,Tohoku University, Sendai, Miyagi
  - Nagano Municipal Hospital, Nagano, Nagano
  - Hokushin Synthesis Hospital, Nakano, Nagano
  - Nagasaki University Graduate School of Biomedical Sciences, Nagasaki, Nagasaki
  - National Hospital Organization Nagasaki Medical Center, Oomura, Nagasaki
  - National Hospital Organization Nagoya Medical Center, Nagoya, Nagoya
  - Nara Medical University Hospital, Kashihara, Nara
  - Niigata Prefectural Cancer Center, Niigata, Niigata
  - Oita Prefectural Hospital, Ōita, Oita Prefecture
  - Kaneda Hospital, Maniwa, Okayama-ken
  - Hospital, University of the Ryukyus, Chutougun, Okinawa
  - Rinku General Medical Center, Izumisano, Osaka
  - Kimen Municipal Hospital, Kimen, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka
  - Osaka City University Graduate School of Medicine, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Sakai Municipal Hospital, Sakai, Osaka
  - Kinki Medical University Hospital, Sayama, Osaka
  - Toyonaka Municipal Hospital, Toyonaka, Osaka
  - Yao Municipal Hospital, Yao, Osaka
  - Saga Medical School Hospital, Saga, Saga-ken
  - Otsu Municipal Hospital, Ōtsu, Shiga
  - Saiseikai Shiga Hospital, Rittō, Shiga
  - Shimane University Faculty of Medicine, Izumo, Shimane
  - Takarazuka City Hospital, Hyōgo, Takarazuka
  - Jichi Medical School Hospital, Shimono, Tochigi
  - Dokkyo University School of Medecine, Shimotsuga, Tochigi
  - Tokushima Red Cross Hospital, Komatsushimachō, Tokushima
  - Tokyo Medical and Dental University Hospital Faculty of Medicine, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku, Tokyo
  - Surugadai Nihon University Hospital, Chiyoda-ku, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Cancer Institute Hospital, Koto-ku, Tokyo
  - Japan Clinical Cancer Research Organization, Koto-ku, Tokyo
  - Showa University Toyosu Hospital, Koto-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - The Jikei University, Minato-ku, Tokyo
  - International University of Health and Welfare Mita Hospital, Minato-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - International Medical Center of Japan, Shinjuku-ku, Tokyo
  - Social Insurange Central General Hospital, Shinjuku-ku, Tokyo
  - Tottori University Faculty of Medicine, Yonago, Tottori
  - Kouseiren Takaoka Hospital, Takaoka, Toyama
  - Yamagata Prefectural Central Hospital, Yamagata, Yamagata
  - Yamanashi Prefectural Central Hospital, Kohfu, Yamanashi

REFERENCES:
- [Derived] Arai H, Takeuchi M, Ichikawa W, Shitara K, Sunakawa Y, Oba K, Koizumi W, Sakata Y, Furukawa H, Yamada Y, Takeuchi M, Fujii M. Correlation of multiple endpoints in the first-line chemotherapy of advanced gastric cancer: Pooled analysis of individual patient data from Japanese Phase III trials. Cancer Med. 2024 Jan;13(1):e6818. doi: 10.1002/cam4.6818. Epub 2023 Dec 23. PMID 38140879
- [Derived] Koizumi W, Kim YH, Fujii M, Kim HK, Imamura H, Lee KH, Hara T, Chung HC, Satoh T, Cho JY, Hosaka H, Tsuji A, Takagane A, Inokuchi M, Tanabe K, Okuno T, Ogura M, Yoshida K, Takeuchi M, Nakajima T; JACCRO and KCSG Study Group. Addition of docetaxel to S-1 without platinum prolongs survival of patients with advanced gastric cancer: a randomized study (START). J Cancer Res Clin Oncol. 2014 Feb;140(2):319-28. doi: 10.1007/s00432-013-1563-5. Epub 2013 Dec 24. PMID 24366758
- [Derived] Fujii M; 0. Chemotherapy for advanced gastric cancer: ongoing phase III study of S-1 alone versus S-1 and docetaxel combination (JACCRO GC03 study). Int J Clin Oncol. 2008 Jun;13(3):201-5. doi: 10.1007/s10147-008-0775-1. Epub 2008 Jun 14. PMID 18553228